CLINICAL TRIAL: NCT01120405
Title: Cardiovascular Safety of Xenon in General Anaesthesia, in Patient With Cardiovascular Risk in Non Cardiac Surgery: A Phase III Multicenter Randomized Controlled Study
Brief Title: Cardiovascular Safety of Xenon in General Anaesthesia, in Patient With Cardiovascular Risk in Non Cardiac Surgery
Acronym: CARVASAXe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Collaborators: Eurofins Biomnis (Other); Monitoring Force Group (Industry); Inferential (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: EudraCT #2010-018703-28
Record Dates: First submitted 2010-05-04; First posted 2010-05-11 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Elevated Cardiac Risk; Coronary Arteries Disease Risk
Keywords: Xenon; Cardiac safety; Cardiovascular risk; Non cardiac surgery; Atherosclerotic vascular surgery
MeSH Terms: interventions — Xenon; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xenon (Experimental): 0.8-1.1 minimum alveolar concentration (MAC) Xenon in 30 % oxygen (Group A)
  Interventions: Drug: Xenon
- sevoflurane (Active Comparator): 0.8-1.1 Minimum Alveolar Concentration (MAC) Sevoflurane in 30 % oxygen (Group B)
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Xenon
  Other Names: LENOXe
  Arms: Xenon
Drug: Sevoflurane
  Other Names: Sevo
  Arms: sevoflurane

SUMMARY:
The Primary Objective is to show non inferiority in cardiac safety (i.e myocardial necrosis-MN- assessed by positive cardiac Troponin I -cTnI- ultrasensitive assay) of a Xenon based general anesthesia procedure in patients with elevated cardiac risk scheduled for atherosclerotic vascular surgery (i.e patient with Coronary Arteries Disease risk) when compared to sevoflurane based general anesthesia procedure, postoperatively up to 3 days.

DETAILED DESCRIPTION:
The Primary endpoint is defined as an increase above the 99th percentile of highly sensitive cardiac Troponin I (cTnI) at any time during the 72 h post operatively. Time frame 3 days post-op;

Key secondary endpoint(s) are routine (Local laboratory) dosage of standard cardiac Troponin I (cTnI) at D1 (24h) and D3 (72 h) post operatively, and also in case of any suspicion of Myocardial Infarction , Routine cardiac safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for atherosclerotic vascular elective surgery with presumed fast-track,
* Cardiac ischaemic risk supported by:

  * History of myocardial infarction older than 1 month and/or
  * Documented Stable angina (asymptomatic ± medical treatment) and/or
  * History of coronary revascularisation, and/or
  * Surgical Risk Index ("Lee" index) ≥ 3.
  * Written informed consent

Exclusion Criteria:

* Unstable angina within the last 30 days,
* Non controlled arterial Hypertension .
* Severe Cardiac heart Failure (NYHA IV)
* Severe Chronic Obstructive Pulmonary Disease
* Patient already randomized in another ongoing clinical trial
* Patient with recent myocardial infarction (M.I) (less than one month )
* Patient already included in a clinical trial
* History of hypersensitivity to study drugs( i.e Xenon, propofol, sevoflurane, desflurane, isoflurane)
* Malignant hyperthermia
* Documented Elevated intracranial pressure
* Preeclampsia or eclampsia
* Pregnancy and lactation
* Presumed uncooperativeness or legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanncik Le Manach, MD, Principal Investigator — CHU PITIE SALPETRIERE, PARIS, FRANCE; Pierre CORIAT, MD Prof, Study Chair — CHU PITIE SALPETRIERE, PARIS, FRANCE; Benoit VALLET, MD Prof, Study Chair — University Hospital, Lille
Locations (13):
- France (13):
  - Nouvel Hopital Civil, Strasbourg, Bas Rhin
  - CHU Nord, Marseille, Bouches du Rhône
  - Centre Hospitalier Universitaire de Caen - Pôle Anesthésie-Réanimation-SAMU, Avenue de la Côte de Nacre, Caen, Calvados
  - CHU Dijon, Dijon, Côte d'Or
  - Hopital Pellegrin, Bordeaux, Gironde
  - CHU Bordeaux Haut Lévèque, Bordeaux, Gironde
  - CHU Rennes, Rennes, Ille et Vilaine
  - CHRU, Hôpital Cardiologique, Département Anesthésie-Réanimation, Bld du Président Jules Leclerc, Lille, Nord
  - Chu Pitie Salpetriere, Paris, Paris
  - Hopital Saint Joseph, Paris, Paris
  - CHU Clermont Ferrand, Clermont-Ferrand, Puy de Dôme
  - Hopital Henri Mondor, Créteil, Val de Marne
  - CHU Poitiers, Service Anesthésie-Réanimation, 2 rue de Milétrie, BP577, Poitiers, Vienne

RESULTS

PARTICIPANT FLOW:
Groups:
- Xenon: 0.8-1.1 Minimum Alveolar Concentration in 30 % oxygen (Group A)
- Sevoflurane: 0.8-1.1 Minimum Alveolar Concentration in 30 % oxygen (Group B)
Period: Overall Study
Arm/Group | Xenon | Sevoflurane
Started | 298 | 302
Completed | 271 | 269
Not Completed | 27 | 33

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): Randomised patients who started general anaesthesia induction. Patients were assigned to the treatment groups as randomised, i.e. the treatment groups were based on the treatment allocated by randomisation.
Groups:
- Xenon: 0.8-1.1 Minimal Alveolar Concentration in 30% oxygen (Group A)
- Sevoflurane: 0.8-1.1 Minimal Alveolar Concentration in 30% oxygen (Group B)
- Total: Total of all reporting groups
Arm/Group | Xenon | Sevoflurane | Total
Number analyzed (Participants) | 295 | 295 | 590
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (10.3) | 71.2 (10.2) | 70.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 52 | 109
  Male | 238 | 243 | 481
Region of Enrollment [Number; unit: participants]
  France | 295 | 295 | 590
Participants with Baseline Cardiac Troponin (Central Laboratory) [Number; unit: participants]
  > 99th percentile | 26 | 26 | 52
  ≤ 99th percentile | 269 | 269 | 538

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Myocardial Necrosis (MN)
Description: Myocardial Necrosis: at least 1 value of serum cardiac troponin I above the 99th percentile (measurement performed by a central laboratory using the ABBOTT-ARCHITECT technique)
Time Frame: 3 Postoperative Days
Population: Per protocol set (PPS): Randomised patients who started general anaesthesia induction and with no major protocol violations. Patients were assigned to the treatment groups as randomised, i.e. the treatment groups were based on the treatment allocated by randomisation.
Measure: Number; unit: participants
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 273 | 261
participants | 57 | 54
Statistical Analysis 1: Comparison: Xenon vs Sevoflurane; The percentage of patients with MN during the 3 postoperative days in the sevoflurane group and in the xenon group was expected to be 20%. The margin of non-inferiority was 10%. Thus the sample size to prove non-inferiority was 252 patients per group with α = 0.025, a power of 0.80 and the following hypotheses: H0: Px-Pc ≥ 10%; H1: Px-Pc < 10%. As it was expected that approximately 15% of patients would be non-evaluable, a total of 600 patients were included; Test type: Non-Inferiority or Equivalence — Non-inferiority of xenon over sevoflurane is accepted if the upper bound of the two-sided 95% CI around the estimated difference is below the prespecified non-inferiority margin of 10%; p = 0.0052, Difference of proportion; Difference of proportion = 0.19, 95% CI 2-sided [-6.70 to 7.07]

2. Secondary Outcome: Number of Participants With Cardiac Troponin I or T Above the 99th Percentile (Local Laboratories)
Description: At least 1 value of serum cardiac troponin I or T above the 99th percentile (measurements performed by local laboratories using different techniques)
Time Frame: 3 Postoperative days
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 295 | 295
participants | 27 [20 to 34] | 25 [20 to 30]
Statistical Analysis 1: Comparison: Xenon vs Sevoflurane; Test type: Superiority or Other; p = 0.7715, Difference of proportion; Difference of proportion = 0.68, 95% CI 2-sided [-3.90 to 5.25]

3. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: Patients with Confirmed Myocardial Infarction (MI) by the Investigators
Time Frame: 3 Postoperative Days
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 295 | 295
participants | 5 [10 to 28] | 3 [10 to 22]
Statistical Analysis 1: Comparison: Xenon vs Sevoflurane; Test type: Superiority or Other; p = 0.4763, Difference of proportion; Difference of proportion = 0.68, 95% CI 2-sided [-1.19 to 2.54]

4. Secondary Outcome: Number of Participants With Cerebro-Vascular Event
Description: Patients with Cerebro-Vascular Event in the FAS
Time Frame: 3 postoperative days
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 295 | 295
participants | 2 | 3
Statistical Analysis 1: Comparison: Xenon vs Sevoflurane; Test type: Superiority or Other; p = 0.6533, Difference of proportion; Difference of proportion = -0.34, 95% CI 2-sided [-1.82 to 1.14]

5. Secondary Outcome: Number of Participants With Life-Threatening Arrhythmia
Description: Patients with Life-Threatening Arrhythmia in the FAS
Time Frame: 3 Postoperative Days
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 295 | 295
participants | 2 | 0
Statistical Analysis 1: Comparison: Xenon vs Sevoflurane; Test type: Superiority or Other; p = 0.1559, Difference of proportion; Difference of proportion = 0.68, 95% CI 2-sided [-0.26 to 1.61]

6. Secondary Outcome: Number of Participants Who Died From Cardiac Origin
Description: No patient died from a cardiac cause during the 3 postoperative days.
Time Frame: 3 postoperative days
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 295 | 295
participants | 0 | 0

7. Secondary Outcome: Number of Participants With Composite Endpoint
Description: Patients with at least 1 event among MN assessed by central laboratory, MI, Cerebro-Vascular event, Life-Threatening Arrhythmia and Death from Cardiac Origin
Time Frame: 3 postoperative days
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 295 | 295
participants | 61 [60 to 62] | 56 [50 to 62]
Statistical Analysis 1: Comparison: Xenon vs Sevoflurane; Test type: Superiority or Other; p = 0.6056, Difference of proportion; Difference of proportion = 1.69, 95% CI 2-sided [-4.74 to 8.13]

8. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: Repeated Systolic Blood Pressure measurements during the perioperative period
Time Frame: From pre-induction to recovery of anesthesia
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 295 | 295
mm Hg
  Baseline | 146.1 (21.6) | 147.3 (23.6)
  Minimum SBP-Induction Time | 90.6 (21.3) | 90.3 (20.7)
  Minimum SBP-Maintenance Time | 94.8 (17.8) | 83.8 (14.2)
  Minimum SBP- Awakening Time | 123.8 (25.1) | 117.6 (23.0)
  Maximum SBP-Induction Time | 156.0 (26.9) | 153.6 (29.6)
  Maximum SBP- Maintenance Time | 157.8 (28.0) | 144.6 (26.1)
  Maximum SBP-Awakening Time | 156.6 (29.1) | 153.4 (27.6)

9. Secondary Outcome: Vital Signs (SBP and DBP Changes)
Description: Changes from baseline for Systolic and Diastolic Blood Pressure (SBP and DBP)
Time Frame: From pre-induction to Postoperative Day 3
Population: Treated set (TS): Randomised patients who received the study medication. Patients were assigned to the treatment groups as treated, i.e. the treatment groups were based on the treatment actually received.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 292 | 294
mm Hg
  SBP-Day 1 | -12.2 (25.4) | -14.2 (26.8)
  SBP-Day 2 | -10.8 (26.6) | -10.7 (25.6)
  SBP-Day 3 | -11.9 (24.7) | -12.2 (25.0)
  DBP-Day 1 | -6.05 (14.91) | -6.15 (15.10)
  DBP- Day 2 | -3.32 (14.53) | -1.46 (13.41)
  DBP-Day 3 | -3.73 (14.05) | -2.61 (13.90)

10. Secondary Outcome: Vital Signs (Heart Rate Changes)
Description: Changes from baseline for Heart Rate (HR)
Time Frame: From pre-induction to Postoperative Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 292 | 294
beats per minute
  HR-Day 1 | 6.35 (12.03) | 6.35 (12.91)
  HR-Day 2 | 8.81 (13.64) | 9.85 (12.93)
  HR-Day 3 | 6.44 (11.72) | 8.90 (14.14)

11. Secondary Outcome: Number of Participants With Chest Pain During the 3 Postoperative Days
Description: Patients with Chest Pain reported at least once per day during the 3 Postoperative Days
Time Frame: From Day 0 until Postoperative Day 3
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 292 | 294
participants
  Day 0 | 0 | 0
  Day 1 | 0 | 2
  Day 2 | 1 | 2
  Day 3 | 2 | 3

12. Secondary Outcome: Urine Output
Description: Urine volume in milliliter (mL) during the first postoperative hours
Time Frame: From Day 0 until Postoperative Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 292 | 294
mL | 1279.0 (723.1) | 1324.4 (631.8)

ADVERSE EVENTS:
Time Frame: Adverse Events observed after the start of study drug administration and during postoperative 3-day period
Description: Participants at risks are the patients from the Treated Set, ie randomised patients who received the study medication.
Arm/Group | Xenon | Sevoflurane
Serious Adverse Events (participants affected / at risk) | 17/292 | 17/294
Other Adverse Events (participants affected / at risk) | 79/292 | 84/294
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xenon (N=292) | Sevoflurane (N=294)
Myocardial Infarction (Cardiac disorders) | 3 | 3
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Subendocardial ischemia (Cardiac disorders) | 0 | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 2 | 3
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 2 | 2
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Operative Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Shunt Trombosis (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 2
Agitation (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Confusional State (Nervous system disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 0 | 1
Troponin Increased (Investigations) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Gallblader Necrosis (Hepatobiliary disorders) | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xenon (N=292) | Sevoflurane (N=294)
Procedural Pain (Injury, poisoning and procedural complications) | 21 | 23
Procedural Hypertension (Injury, poisoning and procedural complications) | 24 | 14
Procedural Nausea (Injury, poisoning and procedural complications) | 21 | 12
Procedural Vomiting (Injury, poisoning and procedural complications) | 16 | 10
Hyperthermia (General disorders) | 13 | 17
Pain (General disorders) | 8 | 15
Hypertension (Vascular disorders) | 17 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Air Liquide Sante International may delay publication or disclosure for a term not exceeding eighteen (18) months with effect from the request in the event that Air Liquide Sante International wishes to seek protection of the results of the Trial by industrial property rights.